CLINICAL TRIAL: NCT06486038
Title: Quatitative MRI of the Spinal Cord in Cervical Myelopathy: Assessment of Microstuctural Damage for Outcome Improvement
Acronym: QCEMY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NEURAD-2022-002
Record Dates: First submitted 2024-06-14; First posted 2024-07-03 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cervical Myelopathy
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidisciplinary and innovative approach (Experimental): MRI examination using experimental sequences on 3 Tesla scanner. Neuromotor assessment by an ad-hoc evaluation of the neuromotor skills that includes upper and lower limb assessment.
  Neurophysiological Assessment: Motor evoked potential (MEP) and Somatosensory evoked potential (SEP) evaluations.
  Neurological and clinical data (including mJOA and Barthel Index) Surgery (if applicable) using a cage in Polyetheretherketone (PEEK) or modern carbon fiber material.
  Interventions: Diagnostic Test: MRI standard and qMRI; Other: MEPs and SSEPs; Other: Neuromotor assessment; Procedure: Anterior cervical discectomy and fusion

INTERVENTIONS:
Diagnostic Test: MRI standard and qMRI — Non-contrast cervical spine MRI including morphological and quantitative MRI sequences on a 3 Tesla scanner. MRI examination includes conventional and experimental sequences
Other: MEPs and SSEPs — Neurophysiological examination by motor and somatosensorial evocked potential using transcranial magnetic stimulation and electrical stimulation to the peripheral nerve
Other: Neuromotor assessment — Upper and Lower limb assessment: Purdue Pegboard Test (PTT), Box and Block test (BBT), Nine Hole Peg Test (NHPT), gait analysis and 30 seconds sit to stand test (30CST)
Procedure: Anterior cervical discectomy and fusion — If applicable: Anterior cervical discectomy and fusion surgery using PEEK or modern carbon fiber material

SUMMARY:
The aim of this low interventional study is to detect microstructural degeneration prior to the presentation, worsening, or persistence following surgical or conservative treatment of cervical degenerative myelopathy signs and symptoms using quantitative imaging metrics and functional biometric analysis.

The endpoints of the study are to collect and compare the clinical, biometric, neurophysiological and imaging data.

The objectives of the study are:

* to implement and validate a novel quantitative Magnetic Resonance (qMRI) protocol clinically for the identification and quantification of microstructural spinal cord damage
* to compare qMRI data to clinical and neuromotor's and corresponding neurophysiological data
* to create an integrated diagnostic tool for early diagnosis and disease monitoring of myelopathy, and for identification of a more reproducible and quantitative scale for assessing reversible and irreversible spinal cord damage combining clinical, biometric, imaging and neurophysiological data in patients suitable for surgical or non-surgical treatment.

Patient will undergo:

* MRI (baseline - 1 month- 6 months)
* clinical data collection (baseline- 1 month - 6 months)
* neuromotor assessment (baseline - 1 month - 6 months)
* neurophysiological assessment (baseline - 6 months)
* surgery if applicable Quantitative MRI of the spinal cord could provide a new objective system for identification of patients who require surgery before developing irreversible clinical damage, and to avoid surgical treatment in those who do not require it. Additionally, quantitative MRI, in combination with clinical data such as, neuromotor tests, could provide an important approach to assess the effectiveness of the therapeutical approach.

DETAILED DESCRIPTION:
Rationale Degenerative cervical myelopathy (DCM) is a common chronic disorder and the most common cause of spinal cord dysfunction in adults, potentially leading to severe functional impairment with high social costs. More than 70% of people younger than 65 years have pathologic or radiologic evidence of cervical degenerative disease. Symptoms of cervical compression develop in about 25% of these people. Consequently, identifying optimal treatment strategies and clinical care pathways for DCM has become a key public health priority. DCM is caused by a progressive deterioration of osseocartilaginous components of the cervical spine leading to a narrowing of the spinal canal and compression of the long tracts and local segmental elements of the Spinal Cord (SC). DCM can lead to progressive disability and paralysis owing to chronic SC compression.

In DCM, an early diagnosis and monitoring are pivotal to avoid or constrain a neurological damage that may persist even after appropriate treatment is provided. Diagnosis of DCM requires agreement between clinical and imaging findings (MRI).

Quantitative MRI of the SC could provide a new objective system for identification of patients who require surgery before developing irreversible clinical damage, and to avoid surgical treatment in those who do not require it. Additionally, quantitative MRI, in combination with clinical data such as, neuromotor tests, could provide an important approach to assess the effectiveness of the therapeutical approach.

The plan with this project is to validate a newer clinically feasible quantitative MRI protocol to depict spinal cord microstructural changes determined by degenerative cervical spine disease, that is highly frequent in the adult population. Investigators are confident that to identify quantitative MRI-derived metrics that could objectively quantify spinal cord damage in degenerative cervical myelopathy, and that could depict microstructural modifications even before neurological signs or signal alterations on morphological MRI sequences are evident. This could be of pivotal importance for more precise indication to surgery and to prevent clinically significant damage that might not be recovered even after surgical treatment. These data will be measured and validated by neurophysiological findings, and compared to current scales and ad-hoc battery of neuromotor skill assessment tests.

Clinical, neurophysiological, biometric and imaging follow-up will be performed to assess the predictive power of the identified metrics.

This study aims to provide a new paradigm for improved depiction of the effects of degenerative cervical spondylosis that could become crucial for an individualized and timely therapeutic decision. In DCM, an early diagnosis is pivotal to avoid neurological damage that may persists even after appropriate treatment is provided. More accurate, integrated clinical, imaging and functional evaluation is also advocated to improve the detection of subtle signs of sensory-motor disturbances, and for increasing the inter-rater and intra-rater reliability of available scales. In the proposed study, for the first time the aim is to: i) integrate T1-based (PSIR, TI-scout) and DTI metrics; ii) compare them to clinical, neurophysiological and neuromotor skill performances, and iii) perform longitudinal pre- and post-operative (ACDF) evaluation.

One important aspect to mention is that this study is performed for the first time, given the availability of the new-generation polyetheretherketone (PEEK) and carbon fiber surgical hardware which allow the acquisition of the advanced quantitative MRI sequences without significant image distortion even when anterior cervical discectomy and fusion (ACDF) is performed.

Through an artificial intelligence approach, investigators also expect to develop a new objective scoring system that will include relevant items from MRI-derived metrics and clinical, neurophysiological and neuromotor skills data. Investigators foresee that the new scoring system could help clinician in identifying patients with the highest risk of progressing to irreversible neurological damage, and that could overcome the limitations of the available clinical scales, that include poor sensitivity and modest inter-rater and intra-rater reliability with limited ability to detect subtle disease progression.

Therefore, the expectation is to identify more objective and sensitive metrics of spinal cord disease burden through the identification of sensitive, objective and quantitative biomarkers of neurological damage in DCM.

The results of this project will provide a new reliable system for identifying patients at risk of progressing to irreversible functional impairment, leading to a patient-centered approach, a cost-effective prevention of neurological deficits, and a cost-effective avoidance of unnecessary surgical interventions.

Objectives

This is a multi-disciplinary study with a focus on subjects affected by cervical spondylosis (DCM) determining several degrees of myelopathy, from mild to severe. The study is aimed at identifying an enhanced clinical, radiological and neuromotor skills evaluation at presentation, seeking to early identify and quantify the disease burden, likely through the depiction and validation of new neuroradiological and functional metrics. This is meant to also tailor and strengthen the indication for surgery, in order to depict microstructural degeneration before signs and symptoms presentation or worsening, since neurological damage may persist even after appropriate treatment has been provided. Additionally, findings from magnetic resonance in combination with neuromotor assessment could be beneficial for patient monitoring after surgery.

Primary objective To implement and validate a novel qMRI protocol clinically for the identification and quantification of microstructural SC damage Secondary objective To compare and correlate clinical and neurophysiological data and detailed movement analysis (overall mobility, walking performance, postural stability, spasticity, upper limb dexterity, detailed movement analysis) with qMRI-derived metrics.

Tertiary objective To elaborate an integrated diagnostic innovative tool for early diagnosis and disease monitoring of myelopathy, and for identification of a more reproducible and quantitative scale for assessing reversible and irreversible spinal cord damage combining clinical, biometric and imaging (qMRI) data assessed at short (1 month) and long-term (6 months) follow-up and neurophysiological data at long-term (6 months) follow-up in patients who underwent either surgical or non-surgical treatment.

The following aims will be pursued to identify more objective and sensitive metrics of the disease burden and prevent the neurological damage from overcoming a clinical threshold.

Primary endpoint Quantitative MRI metrics Secondary endpoint

To combine:

* qMRI data.
* Clinical data (mJOA and Barthel Index).
* Neurophysiologic data (Somatosensory evoked potential (PESS) and Motor evoked potential (MEP)).
* Neuromotor skill assessment (upper and lower limb) Tertiary endpoint Through an artificial intelligence approach above mentioned clinical, biometric, neurophysiological and imaging data assessed at short (1 month) and long-term (6 months) follow-up in patients who underwent either surgical or non-surgical treatment will be combined in order to obtain an enhanced integrated diagnostic powerful tool for early diagnosis and disease monitoring od myelopathy, and for identification of a more reproducible and quantitative scale for assessing reversible and irreversible spinal cord damage.

STUDY POPULATION The propose is a multicentric, prospective, longitudinal study classified as low interventional, enrolling 100 adult subjects with a single-level degenerative spondylosis of the sub-axial cervical spine (C3-C7) as diagnosed on a combination of symptoms, signs and conventional MRI findings.

Patient will undergo:

* MRI (baseline - 1 month- 6 months)
* clinical data collection (baseline- 1 month - 6 months)
* neuromotor assessment (baseline - 1 month - 6 months)
* neurophysiological assessment (baseline - 6 months)
* surgery if applicable The therapeutical treatment would remain standard. No additional imaging sessions will be added in relation to the standard diagnostic and monitoring protocol. Diagnostic MRI will be integrated with advanced sequences which pose no harm for patients and only extend the diagnostic procedure of an interval between 10 and 15 minutes. In addition to traditional practice, patients will receive ad-hoc neuromotor assessment from physical therapists with advanced software for motion analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to give informed consent for participation in the study.
2. Age 18-80.
3. Subjects under evaluation for potential surgical intervention of anterior cervical discectomy and fusion as established by a board-certified neurosurgeon based on clinical and radiological findings according to good clinical practice.
4. Grade I-III single level sub-axial (C3-C7) cervical spinal canal stenosis (Kang, AJR 2011) on a preliminary anatomical MRI.
5. Deficitary or irritative cervical spinal cord symptoms and/or signs in concordance with MRI findings.

Exclusion Criteria:

1. Subjects unable o.r unwilling to give informed consent .
2. Age <18 or > 80
3. Subjects with pacemaker or any other contraindication to undergo high-field (3 Tesla) MRI exam.
4. Pregnancy or planned pregnancy before the end of the study .
5. Co-existing or prior neurological disease of the brain, SC, or peripheral nervous system.
6. Co-existing or prior oncologic disease .
7. Prior surgery in the brain or spine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Novel qMRI protocol clinically for the identification and quantification of microstructural Spinal Cord damage | from baseline until the second follow up (around 6 months)
  A preliminary non-contrast cervical spine MRI including morphological and quantitative sequences on a 3 Tesla scanner:
  * 2D Sagittal T2-w turbo spin-echo (TSE)
  * 2D Sagittal T2-w TSE with short tau inversion recovery (STIR)
  * 3D Sagittal T1-w MP-RAGE with 1x1x1mm3 resolution
  * 2D Transversal T2*-w MEDIC gradient echo
  * 2D Transversal Phase Sensitive Inversion Recovery (PSIR) (0.7x0.7x6.0mm3)
  * 2D Transversal IR TrueFISP sampling 23 different inversion times (TI-scout, 1.0.1.0x10.0mm3)
  * 2D Transversal reduced-FOV ZOOM-EPI spin-echo DTI (180x53mm2 FOV, 5 slices, b=800 s/mm2, 21 directions, 5 interspersed b=0s/mm2 volumes, 0.9x0.9x6.0mm3) with pulse trigger PSIR, TI-scout and DTI sequences will be set perpendicularly to the cord.
  Acquisition of single-slice images at the level of three consecutive intervertebral discs, with the middle one corresponding to the lesion. An image-processing pipeline embedded in a XNAT system will process images.

SECONDARY OUTCOMES:
Integrated diagnostic tool | from month 3 to month 13
  Through an artificial intelligence approach, clinical, biometric, neurophysiological and imaging data assessed at 1 month and 6 months follow-up in patients who underwent either surgical or non-surgical treatment will be combined in order to obtain an enhanced integrated diagnostic powerful tool for early diagnosis and disease monitoring od myelopathy, and for identification of a more reproducible and quantitative scale for assessing reversible and irreversible spinal cord damage.

CONTACTS AND LOCATIONS:
Overall Officials: Letterio S POLITI, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Italy